CLINICAL TRIAL: NCT03914209
Title: Efficacy of a Prophylactic Treatment Using Extended Half-Life (EHL) Clotting Factor for Improving the Musculoskeletal Health of Adult Patients With Hemophilia. Observational Multicenter Study
Brief Title: Extended Half-Life (EHL) Clotting Factor for Improving the Musculoskeletal Health of Patients With Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Other Study IDs: LongHEst
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EHL clotting factor: This study shall not implement any intervention that might alter the normal development of the daily life activities of hemophilia patients included in the study. They will continue with the prophylactic regimen prescribed by their hematologist. Patients will also be asked to continue to develop their physical, work, entertainment and leisure activities in the same way as at baseline.
  Interventions: Other: EHL clotting factor

INTERVENTIONS:
Other: EHL clotting factor — This study shall not implement any intervention that might alter the normal development of the daily life activities of hemophilia patients included in the study. They will continue with the prophylactic regimen prescribed by their hematologist. Patients will also be asked to continue to develop their physical, work, entertainment and leisure activities in the same way as at baseline.

SUMMARY:
Background. Hemophiliac arthropathy is the main long-term physical damage in patients with hemophilia, causing disability and functional limitations.

Objective. Assessment of the efficacy of a prophylactic treatment with EHL products for improving the musculoskeletal health of adult patients with hemophilia.

Study Design. Multicenter observational clinical study. Method. 40 patients with hemophilia A will be included in this study. Patients will be recruited from 5 centers located in various regions of Spain (Community of Madrid, Galicia, Community of Valenciana, Málaga and Vizcaya). The dependent variables will be: bleeding frequency (self-report of bleeding), changes in the dosage of factor VIII with EHL products (rFVIIIFc), pain (measured with the visual analog scale and a pressure Algometer), degree of kinesiophobia (Tampa Scale of Kinesiophobia), degree of adherence to treatment (Veritas-Pro scale), joint health (using the Hemophilia Joint Health Score), muscle strength (using a dynamometer) and functionality (using the 6-Minute Walking Test). Three evaluations will be carried out: baseline, at 6 months, and at the end of the study period, at 12 months. The evolution of quantitative variables shall be analyzed by parametric tests (t-student test) or non-parametric tests (Wilcoxon test). Pearson's correlation coefficient shall be used to obtain the correlation between the dependent and independent variables. By means of a linear regression analysis we will record the percentage influence of the clinical variables relative to the dependent variables measured in this study Expected results. The aim is to establish the effectiveness of the prophylactic treatment in the improvement of the state health, joint pain, muscle strength and functionality in patients with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A
* Patients over 18 years
* Patients under prophylactic treatment with rFVIIIFc concentrates.

Exclusion Criteria:

* Patients with neurological or cognitive disorders preventing the understanding of the various measuring instruments
* Patients who are scheduled for major orthopedic surgery (total arthroplasty)
* Not signed the Informed Consent Document

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size is justified in relation to the prevalence of hemophilia A patients in Spain following prophylactic treatment based on EHL products. Based on the established selection criteria (n = 517, according to the census of the Spanish Federation of Hemophilia), the sample size at the national level would be 146, with a confidence or safety level of 95% and an expected dropout rate of 15%.
  Currently in Spain, treatment with EHL products (rFVIIIFc) in patients with hemophilia A is being implemented and generalized. Thus, for the 8 Spanish regions where the study will be carried out, a sample of 40 patients is established for the work schedule set.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-09-21 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline bleeding frequency after one year of follow-up | Screening visit, at six months and after one year of follow-up
  At baseline, patients will receive a personal self-report of bleeding (hematomas, hemarthrosis and mucous hemorrhagic episodes) where they should indicate the frequency of bleeding during the study period. This record should be delivered to the evaluators in the intermediate assessment and the final evaluation. In this way, changes in the frequency of bleeding throughout the study period will be evaluated

SECONDARY OUTCOMES:
Change from baseline dosage of factor VIII with EHL products after one year of follow-up | Screening visit, at six months and after one year of follow-up
  Changes in the dosage of factor VIII with EHL products (rFVIIIFc) during the study period will be included in all assessments. Dosing data (UI) and weekly administration frequency (days / week) will be collected.
Change from baseline joint pain after one year of follow-up | Screening visit, at six months and after one year of follow-up
  Visual analog scale. This scale will be used to evaluate the perception of joint pain, where joint pain ranges from 0 to 10 points (no pain to maximum perceived pain).
Change from baseline joint pain after one year of follow-up: Pressure algometer | Screening visit, at six months and after one year of follow-up
  Pressure algometer. Measuring instrument used to evaluate pressure joint pain. The instrument shall consist of a measuring device attached to a hard rubber tip 1.1 cm in diameter. Its sphere shall be calibrated in kg/cm2 with divisions of 0.1 kg/cm2. Before taking the measurements, patients will be instructed to say "yes" as soon as pressure exerted by the algometer becomes slightly unpleasant. The pressure algometer shall be kept perpendicular to the surface of the skin with the right hand, stabilizing the axis of the instrument using the thumb and index finger of the left hand. The pressure shall be increased at a uniform rate of approximately 1 kg/cm2 per second. As soon as the subject, according to the instructions, says "yes", the pressure will be stopped and the score will be noted.
Change from baseline kinesiophobia after one year of follow-up | Screening visit, at six months and after one year of follow-up
  Tampa Scale of Kinesiophobia (TSK-11SV). This questionnaire will be used to assess the fear of movement in study patients. It consists of 11 items and the values range from 1 to 4 points (the higher the score, the greater the fear of movement).
Change from baseline joint status after one year of follow-up | Screening visit, at six months and after one year of follow-up
  Hemophilia Joint Health Score (HJHS). This measuring instrument will be used to evaluate the joint condition of knees, ankles, and elbows. It includes 8 items (inflammation and its duration, pain, atrophy and muscle strength, crepitus, and reduced flexion and extension) ranging from 0 to 20 points per joint (the higher the score, the greater the joint deterioration).
Change from baseline lower limb functionality after one year of follow-up | Screening visit, at six months and after one year of follow-up
  6-Minute Walking test (6-MWT). The 6-MWT test is a performance-based test that measures walking speed and the submaximal capacity to perform an exercise. Patients are instructed to walk along a 30 to 50-meter track for 6 minutes attempting to cover as much distance as possible without running. The distance traveled in 6 minutes is recorded, allowing the use of a walking aid or orthopedic devices.
Change from baseline muscle strength after one year of follow-up | Screening visit, at six months and after one year of follow-up
  Dynamometry. The maximum isometric strength of the flexor and extensor muscles of the main joints affected in hemophilia (knees, ankles, and elbows) will be evaluated on both limbs with a manual dynamometer using a mark test. For this test, the rater needs to keep the dynamometer stationary while the patient exerts maximum force against it.
Change from baseline adherence to prophylactic treatment after one year of follow-up | Screening visit, at six months and after one year of follow-up
  Veritas-Pro. Specific adhesion questionnaire for hemophilia patients receiving prophylactic treatment. The Validated Hemophilia Regimen Treatment Adherence Scale - Prophylaxis (Veritas-Pro) questionnaire was developed in the United States and has already been validated in Spanish. The Veritas-Pro scale consists of 24 Likert-type items from 1 to 5, grouped in five dimensions: Time, Dose, Plan, Remembering, Skip and Communicate. The minimum adherence score is 24 points and the maximum adherence score is 120, and in each sub-scale the score ranges from 4 and 20 points.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: No